CLINICAL TRIAL: NCT03555097
Title: Effects of Non-invasive Positive Pressure Ventilation at Different Pressure on Respiratory Mechanics and Neural Respiratory Drive(NRD)in Patients With Stable Chronic Obstructive Pulmonary Disease(COPD)
Brief Title: Effects of Non-invasive Ventilation on Respiratory Mechanics and NRD in Patients With Stable COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-HXNK-010
Record Dates: First submitted 2018-05-31; First posted 2018-06-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2018-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Non-invasive Positive Pressure Ventilation; Respiratory Mechanics; Neural Respiratory Drive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPD Group (Experimental): incremental pressure support
  Interventions: Procedure: incremental pressure support

INTERVENTIONS:
Procedure: incremental pressure support — Inspiratory positive airway pressure (IPAP) gradually increases from 10 to 24 cm water column (cmH2O) with 2 water column (cmH2O) increments. The expiratory positive airway pressure (EPAP) remains 4 water column (cmH2O), and each pressure level is maintained for 5 to 10 minutes.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic respiratory disease characterized by persistent respiratory symptoms and airflow limitation. Pervasive dynamic pulmonary hyperinflation (DPH) and intrinsic positive end-expiratory pressure (PEEPi) can increase inspiratory threshold load and respiratory effort, leading to abnormal changes in respiratory mechanics and neural respiratory drive (NRD). Non-invasive positive pressure ventilation (NPPV) is not only widely used in respiratory failure, but also is one of the important lung rehabilitation strategies. Several studies have reported that the use of biphasic positive airway pressure (BIPAP) mode for NPPV can improve ventilation, reduce NRD, improve NRD coupling, significantly reduce inspiratory muscle load and relieve symptoms. However, relatively few studies are reported that the NPPV is used in COPD patients without non-respiratory failure. Therefore, we suppose that for stable COPD patients without respiratory failure, early intervention with NPPV may reduce DPH, eliminate the adverse effects of PEEPi, reduce the respiratory muscle load, improve the respiratory physiological characteristics, and delay the progression of the disease. Therefore, the purpose of this study is to observe the influence of different levels of BIPAP ventilation on respiratory mechanics and NRD in patients with stable COPD, and to explore whether BiPAP ventilation can be used as a pulmonary rehabilitation method for early intervention of COPD and provide a theoretical basis for subsequent clinical trials.

DETAILED DESCRIPTION:
The patients with COPD will be admitted in one intervention groups. Before using BiPAP ventilation, we will measure the relevant parameters of lung volume, respiratory flow, diaphragm electromyogram, neural respiratory drive mechanical and other baseline index. Then incremental pressure support will be applied to investigate the effects of different levels of BIPAP ventilation on respiratory mechanics and neural respiratory drive.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary function test of forced expiratory volume at one second (FEV1)/forced vital capacity(FVC) < 70% after inhalation of bronchial dilation agent. Patients in a clinically stable state.

Exclusion Criteria:

* Patients they had other respiratory diseases, or evidence of pneumothorax or mediastinal emphysema and pacemaker installed. Patients with acute cardiovascular event and severe cor pulmonale. Patients with poor compliance. An Other causes of diaphragmatic dysfunction.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic function | Change from baseline in diaphragm electromyogram at the pressure of 10cm water column (cmH2O). (5minutes later, 10 minutes later, 15 minutes later, 20 minutes later, 25 minutes later, 30 minutes later, 35 minutes later)
  Diaphragmatic function can be assessed by diaphragm electromyogram (EMGdi), which reflect the physiological activity of the diaphragm and indicate functional status of the central drive.

SECONDARY OUTCOMES:
Respiratory pressure | Change from baseline in diaphragm electromyogram at the pressure of 10cm water column (cmH2O). (5minutes later, 10 minutes later, 15 minutes later, 20 minutes later, 25 minutes later, 30 minutes later, 35 minutes later)
  Respiratory pressure can be assessed by transdiaphragmatic pressure (Pdi).
Respiratory volume | Change from baseline in diaphragm electromyogram at the pressure of 10cm water column (cmH2O). (5minutes later, 10 minutes later, 15 minutes later, 20 minutes later, 25 minutes later, 30 minutes later, 35 minutes later)
  Respiratory volume can be assessed by Tidal volume (VT).
Degree of dyspnea | Change from baseline in diaphragm electromyogram at the pressure of 10cm water column (cmH2O). (5minutes later, 10 minutes later, 15 minutes later, 20 minutes later, 25 minutes later, 30 minutes later, 35 minutes later)
  Difference in the degree of dyspnea can be measured by Borg index.

OTHER OUTCOMES:
Pulse oxygen saturation (SpO2) | Change from baseline in diaphragm electromyogram at the pressure of 10cm water column (cmH2O). (5minutes later, 10 minutes later, 15 minutes later, 20 minutes later, 25 minutes later, 30 minutes later, 35 minutes later)
  Change in SpO2 can be recorded by noninvasive monitoring instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Chen, doctor, Principal Investigator — Zhujiang Hospital,Southern Medical Unversity
Locations (1):
- Zhujiang Hospital,Southern Medical Universicity, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No